CLINICAL TRIAL: NCT02093533
Title: EVALUATING THE MORPHOFUNCTIONAL EFFECTS OF ECULIZUMAB THERAPY IN PRIMARY MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS: A PILOT, SINGLE ARM STUDY IN TEN PATIENTS WITH PERSISTENT HEAVY PROTEINURIA
Brief Title: Eculizumab in Primary MPGN
Acronym: EAGLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Alexion Pharma Italy s.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAGLE; 2013-003826-10 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Membranoproliferative Glomerulonephritis
Keywords: Membranoproliferative glomerulonephritis; Nephrotic syndrome; Proteinuria; Alternative complement pathway; Complement inhibition; Eculizumab
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative; Nephrotic Syndrome; Proteinuria | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eculizumab (Experimental): Patient Body weight ≥40 kg: initial phase 900 mg weekly x 4 and maintenance phase 1200 mg at week 5; then 1200 mg every 2 weeks Patient Body weight 30 - <40 kg : initial phase 600 mg weekly x 2 and maintenance phase 900 mg at week 3; then 900 mg every 2 weeks
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab
  Other Names: Soliris

SUMMARY:
Membranoproliferative glomerulonephritis (MPGN) is the third or fourth leading cause of end stage renal disease among the primary glomerulonephritis. Hyperactivation of the alternative complement pathway and familial forms for all types of MPGN have been reported suggesting that genetic abnormalities may play a predisposing role to the disease. In recent case reports Eculizumab, a monoclonal antibody that binds to C5 to prevent formation of the membrane attack complex ,is a safe and effective therapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven primary MPGN
* Creatinine clearance >20 ml/min per 1.73m2
* 24-hour proteinuria persistently exceeding 3,5g in adults or exceeding 40mg/h/m2 in children (or exceeding 2mg protein/mg creatinine in children spot urine samples)
* Persistently low C3 levels in at least two consecutive evaluations
* Persistently high sC5b9 levels (>1000 ng/ml) in at least two previous consecutive evaluations
* Written informed consent (by parents or tutors if underage)

Exclusion Criteria:

* Age ≥75 years
* Secondary MPGN (evidence of infection, immunological disease including vasculitis, systemic diseases and proliferative disorders)
* Evidence at kidney biopsy evaluation of severe chronic histological changes that very unlikely could benefit of eculizumab therapy
* Concomitant steroid or immunosuppressive therapy for immuno-mediated disease
* Pregnancy or lactating
* Childbearing potential without effective contraception
* Any clinically relevant condition that might affect completion of the study participation and/or confound study results
* Inability to understand the potential risks and benefits of the study
* Legal incapacity

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
24hours proteinuria | Changes from baseline at week 1,12,24,36,48 and 72.

SECONDARY OUTCOMES:
Terminal complement complex (sC5b-9) levels | Changes from baseline at 1,2, 3, 4,12,24,36,48,52,56,60 and 72 week.
Glomerular filtration rate (GFR) measured by iohexol plasma clearance and estimated. | Changes from Baseline at 1,24, 48 and 72 week.
Time to disease progression. | Up 72 week.

OTHER OUTCOMES:
Number of participants with Adverse Events as a measure of safety. | Participants will be followed for the duration of the study, an expected average of 72 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Ospedale Pediatrico "Giovanni XXIII" - U:O Nefrologia, Bari, BA
  - A.O. Papa Giovanni XXIII - U.O. Nefrologia e Dialisi/IRCCS IRFMN - Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò, Bergamo, BG
  - Policlinico Sant'Orsola -Malpighi - U.O.S. Nefrologia e dialisi pediatrica, Bologna, BO
  - Policlinico "G.Martino" - U.O. Nefrologia e Dialisi, Messina, ME
  - Policlinico Universitario di Padova - U.O. Nefrologia Pediatrica, Padua, PD
  - Ospedale Centrale, Bolzano
  - Policlinico "Federico II" - U.O. Nefrologia, Napoli
  - Ospedale degli Infermi - U.O. Nefrologia e Dialisi, Rimini
  - C.I. Columbus-Università Cattolica del S.Cuore - UOC Nefrologia e Dialisi, Roma
  - Ospedale Pediatrico "Bambin Gesù" - U.O. Nefrologia, Roma
  - Presidio Ospedaliero O.I.R.M. "Sant'Anna" - U.O. Nefrologia, Torino
  - Ospedale "Santa Chiara" - U.O. Nefrologia, Trento
  - Ospedale Cà Foncello - U.O. Nefrologia, Treviso